CLINICAL TRIAL: NCT04496843
Title: Validation of the Diagnostic Performance of the Sleep Apnea Syndrome by the Withings HWA09 Device
Acronym: VPASH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Withings (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-A01347-50
Record Dates: First submitted 2020-07-27; First posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients referred for an overnight in-lab PSG: Simultaneous assessment of SAS with Withings HWA09 Device and overnight PSG
  Interventions: Diagnostic Test: HWA09 Measurement

INTERVENTIONS:
Diagnostic Test: HWA09 Measurement — Simultaneous recording of Withings HWA09 Device and PSG devices for the reference.

SUMMARY:
Sleep Apnea Syndrome (SAS) is a common pathology affecting between 4 and 8% of the general population. It aggravates morbidity and cardio-metabolic mortality and is responsible for accidents related to vigilance disorders. It is estimated that 80%% of SAS cases are not diagnosed and therefore not treated. It is however impracticable to propose a diagnostic test of polygraphy (PG) or polysomnography (PSG) to every patient because of the cost and insufficient availability of these exams. It would therefore be useful to carry out a screening test before directing the patient to a complete test.

Several simplified polygraph systems with 2 or 3 channels have been proposed (nasal cannula, oximetry, heart rate) but they generally record only one night and remain intrusive enough to perturb the sleep.

The Withings HWA09 is a wrist-worn watch, which allows screening of SAS from four signals: movement, heart rate, breathing rate and blood oxygen saturation (SpO2). The objective of the present study is to validate the diagnostic performance of the Withings HWA09 for the detection of SAS compared to PSG.

DETAILED DESCRIPTION:
Subjects are patients having a prescription for a one-night polysomnographic consultation in order to diagnose potential sleep disorders. The investigator will collect the consent before including any patient in this study. The study last one night per patient, during which saturation signal recordings and the sleep apnea detection will be made by the HWA09 watch, in comparison to the polysomnography.

ELIGIBILITY:
Inclusion Criteria:

* Adults, men and women, between 18 and 70 y/o
* Patient addressed for a polysomnography because of a suspicion of sleep respiratory disorders
* Subject having expressed his/her consent to take part in the study

Exclusion Criteria:

* Recording under continuous positive pressure
* Subject having refuse to give his/her consent
* Vulnerable subjects according to regulation in force :
* Pregnant, parturient or breastfeeding women
* Subjects having a known allergy to one of the components of the sensor (silicon, stainless steel, sapphire glass)
* Subjects deprived of liberty by a court, medical or administrative order
* Subjects legally protected or unable to express their non-opposition to take part in the study
* Subjects unable to express their consent due to linguistic or mental incapacities

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients referred for an in-lab polysomnography
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2020-01-16 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of Withings HWA09 at AHI threshold value of 5/h in PSG | 1 year
  Sensitivity and specificity for SAS detection by Withings HWA09 compared to PSG at apnea-hypopnea index (AHI) threshold value of 5/h in PSG.
Sensitivity and Specificity of Withings HWA09 at AHI threshold value of 15/h in PSG | 1 year
  Sensitivity and specificity for SAS detection by Withings HWA09 compared to PSG at AHI threshold value of 15/h in PSG.
Sensitivity and Specificity of Withings HWA09 at AHI threshold value of 30/h in PSG | 1 year
  Sensitivity and specificity for SAS detection by Withings HWA09 compared to PSG at AHI threshold value of 30/h in PSG.

SECONDARY OUTCOMES:
Sensitivity and Specificity of the desaturation detected by Withings HWA09 | 1 year
  Sensitivity and specificity of the desaturation detection by Withings HWA09 compared to an oximeter with the Oxygen Desaturation Index (ODI)
Accuracy of Withings HWA09 to estimate total sleep time (TST) given by PSG | 1 year
  Bias and mean absolute error (MAE)
Impact of the proportion of apnea events on the performance of Withings HWA09 | 1 year
  Bias and MAE for apnea index (AI) estimated by Withings HWA09 compared to PSG results
Impact of the proportion of hypopnea events on the performance of Withings HWA09 | 1 year
  Bias and MAE for hypopnea index (HI) estimated by Withings HWA09 compared to PSG results
Influence of the position of the sleeper (supine vs prone/lateral decubitus position) on the error of the AHI predicted by Withings HWA09 compared with PSG | 1 year
  Average difference of AHI between Withings HWA09 and the PSG in each position
Reliability of Withings HWA09 | 1 year
  Rate of unusable of lost nights

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Roisman, Principal Investigator — Antoine Béclère Hospital
Locations (2):
- St Pierre Hospital, Brussels, Belgium
- Antoine Béclère Hospital, Clamart, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No